CLINICAL TRIAL: NCT03095196
Title: Multipolar Pacing by Cardiac Resynchronization Therapy With a Defibrillator as Treatment in Type 2 Diabetes Mellitus Failing Heart Patients: Impact on Responders Rate, and Clinical Outcomes.
Brief Title: Multipolar CRT-d and Diabetes
Status: Completed | Type: Observational
Sponsor: Celestino Sardu (Other)
Responsible Party: Sponsor-Investigator, Celestino Sardu, Clinical professor, University of Campania Luigi Vanvitelli
Organization: University of Campania Luigi Vanvitelli (Other)
Other Study IDs: JPS912.915
Record Dates: First submitted 2017-03-09; First posted 2017-03-29 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Diabetes; Heart Failure; Heart Failure NYHA Class II; Heart Failure NYHA Class III
MeSH Terms: conditions — Diabetes Mellitus; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- T2DM, treated by multipolar CRT-d: Type 2 diabetes (T2DM) affected by heart failure (HF), treated by multipolar CRT-d, plus maximal drug therapy.
  Interventions: Device: Multipolar CRT-d, plus conventional drug therapy for HF.; Drug: HF drugs
- T2DM, treated by bipolar CRT-d: Type 2 diabetes (T2DM) affected by heart failure (HF), treated by bipolar CRT-d, plus maximal drug therapy.
  Interventions: Device: Bipolar CRT-d, plus conventional drug therapy for HF.; Drug: HF drugs

INTERVENTIONS:
Device: Multipolar CRT-d, plus conventional drug therapy for HF. — A random CRT-d implant performed via multipolar left ventricle lead, in failing heart patients treated by maximal drug therapy.
  Groups: T2DM, treated by multipolar CRT-d
Device: Bipolar CRT-d, plus conventional drug therapy for HF. — A random CRT-d implant performed via bipolar left ventricle lead (group B), in failing heart patients treated by maximal drug therapy.
  Groups: T2DM, treated by bipolar CRT-d
Drug: HF drugs — full medical therapy to treat HF symptoms and its progression.

SUMMARY:
Background: Type 2 Diabetes Mellitus (T2DM) is a multi factorial disease, affecting clinical outcomes in failing heart (HF) patients treated by Cardiac Resynchronization Therapy with a defibrillator (CRT-d).

Methods: One hundred and ninety five T2DM patients will receive a CRT-d treatment. Randomly the study population will receive a CRT-d via multipolar left ventricle (LV) lead pacing (n 99 as Multipolar group), v/s a CRT-d via bipolar LV pacing (n 96, as Bipolar group). These patients will be followed by clinical, and instrumental assessment, and telemetric device control at follow up. Study design will be to evaluate, in failing heart T2DM patients, cardiac deaths, all cause deaths, arrhythmic events, CRT-d responders rate, hospitalizations for HF worsening, phrenic nerve stimulation (PNS), and LV catheter dislodgment events (and re-intervention for LV catheter re-positioning), comparing multipolar CRT-d v/s bipolar CRT-d group of patients at follow up.

DETAILED DESCRIPTION:
Introduction: Type 2 diabetes mellitus (T2DM) is a worldwide increasing disease, impacting on heart functions, and cardiac diseases, and outcomes. T2DM may lead to heart failure (HF) disease, and conditioning HF disease progression, and the response to treatments. In HF patients, cardiac resynchronization therapy with a defibrillator (CRT-d) is a well-established treatment to improve symptoms, quality of life, NYHA class, and clinical outcomes. T2DM may condition the CRT-d response. The advancement of CRT-d technology worked to reduce implant complications, phrenic nerve stimulation (PNS) events, and left ventricle (LV) catheter dislodgments, and to ameliorate the CRT-d responders rate, and clinical outcomes. The multipolar LV lead pacing represented one of the waited technological advancement in CRT-d technology, resulted in a stable and continuous CRT-d pacing. The stable and continuous CRT-d pacing may condition the prognosis, and CRT-d responders rate in failing heart patients. At our knowledge, there are not data investigating these effects in a population of T2DM failing heart subjects. In this study T2DM failing heart patients randomly received a CRT-d via multipolar LV lead and/or a CRT-d via bipolar LV lead. In these patients we evaluated, as primary study endpoints, PNS events, LV lead dislodgments, interventions for LV re-positioning, cardiac deaths, all cause deaths, stroke events, and hospitalizations for HF worsening. As secondary endpoints we evaluated arrhythmic events, strokes, and CRT-d responders rate. Our study hypothesis was that, in T2DM failing heart patients multipolar LV pacing may lead to a reduction of PNS episodes, LV leads dislodgments, and interventions to re-positioning LV leads, leading to a significant amelioration of the HF clinical status, and of the CRT-d responders rate. These effects induced by multipolar CRT-d pacing may reduce arrhythmic events, hospitalizations for HF worsening, and of cardiac deaths, and all cause deaths in T2DM patients.

Methods: From September 2012 to September 2015 we conducted a multicenter, prospective, randomized study at University of Campania Luigi Vanvitelli, Italy, Catholic University of Sacred Heart, Campobasso, Italy, and John Paul II Research and Care Foundation, Campobasso, Italy. We screened 213 consecutive T2DM patients with stable chronic HF, NYHA functional class II or III, left bundle branch block, severe left ventricle ejection fraction reduction (LVEF < 35%), stable sinus rhythm, candidates to receive a CRT-d treatment according to the international guidelines. Exclusion criteria were: age <18 or >75 years, ejection fraction >35%, previous implantable cardioverter defibrillator (ICD), CRT-d and/or pacemaker implant, absence of informed patient consent, and any condition that would make survival for 1 year unlikely. 198 eligible patients were included in the study, and received a CRT-d treatment, and a traditional CRT-d ambulatory monitoring. The CRT-d has randomly undergone via multipolar left lead pacing (n 101) v/s bipolar left lead pacing (n 98). Study population was divided in Multipolar CRT-d group (multipolar LV pacing), v/s Bipolar CRT-d group (bipolar LV pacing), according to the LV lead stimulation catheter used, and implanted at enrolment. 99 patients in Multipolar CRT group v/s 96 patients in the Bipolar CRT group completed the follow up. All patients were informed about the study nature, and gave their written informed, and signed consent to participate in the study.

Study protocol: 199 patients received a CRT-d, then divided in multipolar CRT-d patients (n 101), and bipolar CRT-d patients (n 98). Before interventions, baseline laboratory studies, including HbA1c, lipid panel, and fibrinogen, were determined. Follow-up was concluded at 12 months after CRT-d implant. Responders patients to a CRT-d treatment were defined by evidence of LV reverse remodeling, 6 minutes-walk improvement and Minnesota Living with Heart Failure scale improvement. Enrolled patients were followed by clinical, instrumental assessment, and device telemetric control at follow up. During these visits we reported lead functionality parameters, and arrhythmic events in CRT-d recipients, PNS episodes, and CRT-d effect on clinical outcomes. This study was conducted from September 2012 to December 2015. The study was conducted in accordance with the Declaration of Helsinki. The Ethics Committees of all participating institutions approved the protocol.

Intervention phase: CRT-d implant procedure, and LV pacing leads positioning Experienced electrophysiologists performed CRT implant procedures, that were standardized. Right atrial catheters were all placed in right atrial appendage, right ventricular catheters in right ventricle apex, as indicated by antero-posterior, right anterior, and left anterior oblique views projections at radioscopic imaging. LV epicardial catheters were placed by percutaneous coronary sinus catheterization. In this case we have chosen, by previous described radioscopic projections and angiography, a lateral and/or posterior-lateral target vessel, according to international guidelines recommendations. We randomly chose a multipolar and/or a bipolar left ventricle pacing lead, as described before in the text. Implantation duration was defined as the time between skin incision until suture. Measurements were repeated within 24hours of implantation using the implanted pulse generator and pacemaker programmer, and then 10th days, 6th month, 12th month after discharge at follow up. The sensing and pacing LV configurations were defined by 10 bipolar configurations for multipolar LV pacing modality, and at least 4 different left ventricle pacing configurations (LV tip to either LV ring or right ventricular (RV) coil, and LV ring to either LV tip or RV coil) for the bipolar left ventricle pacing group. LV pacing leads were connected to an appropriate bipolar CRT-D device.

Follow up phase:

Lead functionality parameters Right atrium, right ventricle, and left ventricle leads functionality parameters were measured, as P, and R-wave amplitude values (sensing thresholds), lead impedances values (impedance thresholds), and lead pacing outputs values (pacing thresholds). The sensing thresholds values were obtained from the intra-cardiac electrograms records, measured using a sensing configuration. The pacing thresholds, and impedance thresholds values, were measured using pacing catheter configurations. To measure intra thoracic impedance (Ohm), and pacing thresholds (Volt for milliseconds), we focused on the right ventricle (RV) coil electrode to device case pathway configuration, and on the left ventricle (LV) tip to LV ring configuration. These parameters were evaluated during ambulatory follow up visits, and device interrogations at follow up.

Arrhythmic events in CRT-d recipients Arrhythmic events were defined as atrial fibrillation (AF), ventricular tachycardia (VT), and ventricular fibrillation (VF) episodes, and implantable cardioverter defibrillator (ICD) shocks. AF was defined as paroxysmal, and/or not paroxysmal according to authors suggestions. VT was defined as arrhythmia originating from ventricular chambers, sustained and/or not sustained by arrhythmic event duration. VF was defined as a fibrillating arrhythmia originating from ventricular chambers, and associated to hemodynamic instability, and cardiac arrest. By CRT-d devices interrogations at follow up we reported ICDs shocks for each CRT-d patient, at 10th days, 6th month, and at 12th month after implantation.

Phrenic nerve stimulation events PNS and left ventricle pacing leads threshold were measured by a standard protocol at CRT-d implant, and during all follow up durations by CRT-d devices interrogations. In case of PNS diagnosis during follow up, by patients symptoms assessment, devices interrogations, and physician ambulatory diagnosis, we reached the best left ventricle lead pacing configuration to solve PNS.

LV leads dislodgments LV catheter dislodgments resulted by the movement of the catheter into and out of the coronary sinus implantation vessel site, and then causing a change in the catheter tip location. It was diagnosed by patients clinical symptoms, hospital admissions schedules, hospital discharge schedules, and during medical interrogation at follow up visits, and was confirmed by radiographic biplane projections assessment.

CRT-d effect on clinical outcomes CRT-d responders rate was evaluated by periodic clinical examination, and echocardiography assessment. Interventions for LV lead re-positioning were defined as interventions done after the first CRT-d implant, and were evaluated by hospital admissions schedules, hospital discharge schedules, and medical interrogation at follow up visits. These interventions were done in case of LV catheter dislodgments. Hospitalization rate was reported during telephonic interviews, by hospital admissions schedules, hospital discharge schedules, and during medical interrogation at follow up visits. Cardiac deaths, all cause of deaths, and stroke events were evaluated during office follow up visits 10 days after clinical discharge, and after 6th and 12th months by the treating physician, by telephonic interview, hospital admission, and discharge schedules. At each clinical follow-up, right atrial, right ventricular, and left ventricular leads functionality, atrial, and ventricular arrhythmias, ICD shocks, and biventricular pacing percentage, were evaluated and reported for each patient. NYHA classification was re-assessed, and patients graded their overall condition as unchanged or slightly, moderately, or markedly worsened, or improved since randomization by global self-assessment. All patients were instructed to report about devices alarms, loss of lead capture, phrenic nerve stimulation, and arrhythmias. All patients were instructed regularly to assess body weight, occurrence of dyspnea, and any clinical symptom. At each visit patients were asked whether medical events or symptoms suggestive of cardiac arrhythmias occurred, and an ECG, and an ECG Holter monitoring, were both performed to detect the presence of asymptomatic arrhythmias. Clinical evaluations included physical examination, vital signs, and review of adverse events.

Study endpoints As primary endpoints we monitored CRT-d effect in multipolar CRT-d patients v/s bipolar CRT-d patients in terms of PNS, LV leads dislodgments, interventions to re-position LV leads, hospitalization rate for HF worsening, cardiac deaths, and all cause deaths. As secondary endpoints we monitored CRT-d responders rate, arrhythmic events, and strokes in both groups (multipolar CRT-d v/s bipolar CRT-d patients).

Statistical methods A qualified statistician analyzed all collected data. The patients were divided before in multipolar CRT-d group v/s bipolar CRT-d group, and during follow up visits, and controls in CRT-d responders v/s CRT-d non-responders. Continuous variables were expressed as means and standard deviations, and were tested by two-tailed Student t test for paired or unpaired data, as appropriate, or by one-way analysis of variance (ANOVA) for more than two independent groups of data. The categorical variables were compared by chi-square or Fisher exact test where appropriate. Survival analysis was performed with the use of the Kaplan-Meier method. Predictors of the study endpoints were evaluated by using Cox regression models in which covariates for the adjustment were selected if associated with a p value ≤0.25 at univariate analysis. A stepwise method with backward elimination was used and hazard ratios (HR) with 95% confidence intervals (CI) were derived. We considered a two-sided p value of less than 0.05 as statistically significant. The statistical analysis was performed using the SPSS software package for Windows 17.0 (SPSS Inc., Chicago Illinois).

ELIGIBILITY:
Inclusion Criteria:

T2DM patients with stable chronic heart failure, New York Heart Association (NYHA) functional class II or III, left bundle branch block, severe left ventricle ejection fraction reduction (LVEF < 35%), stable sinus rhythm, candidates to receive a CRT-d treatment

Exclusion Criteria:

age <18 or >75 years, ejection fraction >35%, previous implantable cardioverter defibrillator (ICD), CRT-d and/or pacemaker implant, absence of informed patient consent, and any condition that would make survival for 1 year unlikely.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 213 consecutive T2DM patients with stable chronic heart failure, New York Heart Association (NYHA) functional class II or III, left bundle branch block, severe left ventricle ejection fraction reduction (LVEF < 35%), stable sinus rhythm, candidates to receive a CRT-d treatment according to the international guidelines. Exclusion criteria were as follows: age <18 or >75 years, ejection fraction >35%, previous implantable cardioverter defibrillator (ICD), CRT-d and/or pacemaker implant, absence of informed patient consent, and any condition that would make survival for 1 year unlikely.
Sampling Method: Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2014-09-01 (Actual); Study Completion 2015-09-01 (Actual)

PRIMARY OUTCOMES:
Phrenic nerve stimulation episodes | 24 months
  As primary endpoints we monitored CRT-d effect in multipolar CRT-d patients v/s bipolar CRT-d in terms of Phrenic nerve stimulation episodes (PNS). PNS were assessed by left ventricle pacing leads threshold by a standard protocol at CRT-d implant, and during all follow up durations by CRT-d devices interrogations. In case of PNS diagnosis during follow up, by patients symptoms assessment (phrenic simulations during CRTd pacing), and confirmed by devices interrogations, and physician ambulatory diagnosis, we reached the best left ventricle lead pacing configuration to solve PNS.
Left Ventricle (LV) leads dislodgments | 24 months
  As primary endpoints we monitored CRT-d effect in multipolar CRT-d patients v/s bipolar CRT-d in terms of LV leads dislodgments, as confirmed by the movement of the catheter into and out of the coronary sinus implantation vessel site, and then causing a change in the catheter tip location. It was diagnosed by patients clinical symptoms, hospital admissions schedules, hospital discharge schedules, and during medical interrogation at follow up visits, and was confirmed by radiographic biplane projections assessment.
Interventions to re-position LV leads | 24 months
  As primary endpoints we monitored CRT-d effect in multipolar CRT-d patients v/s bipolar CRT-d in terms of interventions done after the first CRT-d implant to re-position LV leads in case of LV leads dislodgments. This endpoint was evaluated by hospital admissions schedules, hospital discharge schedules, and medical interrogations at follow up visits. These interventions were done in case of LV catheter dislodgments.
Hospitalization rate for HF worsening | 24 months
  As primary endpoints we monitored CRT-d effect in multipolar CRT-d patients v/s bipolar CRT-d in terms of hospitalization rate for HF worsening. Hospitalization rate was reported during telephonic interviews, by hospital admissions schedules, hospital discharge schedules, and during medical interrogation at follow up visits.
Cardiac deaths | 24 months
  As primary endpoints we monitored CRT-d effect in multipolar CRT-d patients v/s bipolar CRT-d in terms of Cardiac deaths. Cardiac deaths were evaluated during office follow up visits 10 days after clinical discharge, and after 6th and 12th months by the treating physician, by telephonic interview, hospital admission, and discharge schedules.
All cause deaths. | 24 months
  As primary endpoints we monitored CRT-d effect in multipolar CRT-d patients v/s bipolar CRT-d in terms of all cause deaths. Alla cause deaths were evaluated during office follow up visits 10 days after clinical discharge, and after 6th and 12th months by the treating physician, by telephonic interview, hospital admission, and discharge schedules.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sardu C, Barbieri M, Santamaria M, Giordano V, Sacra C, Paolisso P, Spirito A, Marfella R, Paolisso G, Rizzo MR. Multipolar pacing by cardiac resynchronization therapy with a defibrillators treatment in type 2 diabetes mellitus failing heart patients: impact on responders rate, and clinical outcomes. Cardiovasc Diabetol. 2017 Jun 9;16(1):75. doi: 10.1186/s12933-017-0554-2. PMID 28599667